CLINICAL TRIAL: NCT00289978
Title: A 24-month, Double-blind, Randomized, Multicenter, Placebo-controlled, Parallel-group Study Comparing the Efficacy and Safety of Fingolimod 1.25 mg and 0.5 mg Administered Orally Once Daily Versus Placebo in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Efficacy and Safety of Fingolimod in Patients With Relapsing-remitting Multiple Sclerosis
Acronym: FREEDOMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CFTY720D2301
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Results first posted 2011-03-16 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; FTY720; Fingolimod
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Fingolimod 1.25 mg (Experimental)
  Interventions: Drug: Fingolimod 1.25 mg
- Fingolimod 0.5 mg (Experimental)
  Interventions: Drug: Fingolimod 0.5 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fingolimod 1.25 mg — Patients self-administered fingolimod 1.25 mg capsules orally once daily.
  Arms: Fingolimod 1.25 mg
Drug: Fingolimod 0.5 mg — Patients self-administered fingolimod 0.5 mg capsules orally once daily.
  Arms: Fingolimod 0.5 mg
Drug: Placebo — Patients self-administered a fingolimod placebo capsule orally once daily.
  Arms: Placebo

SUMMARY:
This study assessed the efficacy, safety, and tolerability of 2 doses of oral fingolimod (1.25 mg/day and 0.5 mg/day) compared to placebo in patients with relapsing-remitting multiple sclerosis (RRMS)

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between ages 18-55 with a diagnosis of multiple sclerosis
* Patients with a relapsing-remitting disease course
* Patients with EDSS score of 0-5.5

Exclusion Criteria:

* Patients with other chronic disease of the immune system, malignancies, acute pulmonary disease, cardiac failure, etc.
* Pregnant or nursing women

Other protocol-defined inclusion/exclusion criteria applied to this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1272 (Actual)
Dates: Start 2006-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (112):
- Australia (5):
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - North Gosford Private Hospital, Burrabil Avenue, Suite 17, Gosford
  - Strategic Health Evaluators, Chatswood
  - St Vincent's Hospital Melbourne, Department of Clinical Neurosciences, Fitzroy
  - Austin Health, Department of Neurology, Heidelberg
- Belgium (8):
  - Algemeen Ziekenhuis St. Jan, Department of Neurology, Ruddershove, Brugge
  - Erasme Hospital, Route de Lennik 808, Brussels Capital
  - CHU Charleroi, Hôpital Civil, Boulevard Paul Janson 92, Charleroi
  - University Hospital Gasthuisberg, Department Neurology, Herestraat 49, Leuven
  - AZ Alma, Department of Neurology & Rehab-Umit, Gentsesteenweg 132, Sijsele
  - Regionaal Ziekenhuis, St.Trudo, Diestersteenweg 100,, St.Truiden
  - MS Klinik, Boemerangstraat 2, Overpelt
  - National Multiple Sclerose Centrum v.z.w, Vanheylenstraat 16, Melsbroek
- Canada (8):
  - University of British Columbia, Me498 2211 Wesbrook Mall, Vancouver, British Columbia
  - DMSRU - Capital Health, Halifax, Nova Scotia
  - Kingston General Hospital, MS Clinic, Connell 7, 76 Stuart Street, Kingston, Ontario
  - Nepean Medical Center, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Clinical Trials Office,, Trillium Health Center, 00 Queesway West, Mississauga, Ontario
  - Hopital Maisonneuve-Rosemont, Recherche Clinique de Neurologie, Montreal, Quebec
  - University of Saskatchewan, Regina, Saskatchewan
- Czechia (11):
  - Military Hospital of Brno, Department of Neurology, Zabrdovicka 3, Brno
  - Faculty Hospital St. Anne, First Department of Neurology, Pekarska 53, Brno
  - Faculty Hospital, Department of Neurology, I.P. Paulova 6, Olomouc
  - Hospital of Pardubice, Department of Neurology, Kyjevska 44, Pardubice
  - Faculty Hospital, Department of Neurology, Alej Svobody 80, Plzeň
  - Neurologicka klinika, Fakultni nemocnice, Kralovske Vinohrady, Srobarova 50, Prague
  - Faculty Hospital Motol, MS Center, Department of Neurology, V Uvalu 84, Prague 5
  - Vseobecna fakultni nemocnice, MS Centrum, Neurologicka Klinika, Karlovo Namesti 32, Praha 2
  - MS Centrum, Neurology Department of Hospital Teplice, Duchcovska 53, Teplice
  - Centrum neurologicke pece, Jiraskova 1389, Rychnov Nad Kneznou
  - Facultní Nemocnice Spoliklinikou Ostrava, Neurology Department, Ostrava
- Finland (5):
  - Helsinki Headache Center Postitalon Lääkäriasema, Mannnerheiminaukio 1 B 2 Floor, Helsinki
  - Finnish Special Neurology Center Ltd., Brahenkatu 11 D,, Turku
  - Suomen Terveystalo/ Päänsärkykeskus, Tampere, Hämeenkatu 18, 6th Fl., Tampere
  - Turku University Hospital, Neurology Department 799, Kiinanmyllynkatu 11- 14, Turku
  - Hyvinkään sairaala, Neurologian Poliklinikka, Sairaalankatu 1, Hyvinkää
- CHU La Timone, Service Neurologie, Boulevard Jean Moulin, Marsielle Cedex 5, France
- Germany (13):
  - Investigational Site, Berlin
  - Investigational Site, Düsseldorf
  - Investigational Site, Giessen
  - Investigational Site, Hamburg
  - Investigational Site, Leipzig
  - Investigational Site, Magdeburg
  - Investigational Site, München
  - Investigational Site, Münster
  - Investigational Site, Regensburg
  - Investigational Site, Seesen/Harz
  - Investigational Site, Stuttgart
  - Investigational Site, Tübingen
  - Investigational Site, Würzburg
- Greece (4):
  - Athens Naval Hospital, Neurology Department, Athens
  - Neurology Department Athens General Hospital, G. Gennimatas, Mesogeion 154 Ave., Athens
  - 1st IKA Papadimitriou Neurology Dept, Terma Zaimi, Melissia-Athens
  - University General Hospital of Thessaloniki "AHEPA", B' University Department of Neurology, Thessaloniki
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Carmel Medical Center, Haifa
  - Sieff Medical Center, Safed
  - Sheba - Medical Center, Tel Hashomer, Ramat-Gan,
- Kaunas University Hospital Department of Neurology, Eiveniu 2, Kaunas, Lithuania
- Netherlands (6):
  - Academisch Ziekenhuis VU, De Boelelaan 1118, Amsterdam
  - St. Antonius Ziekenhuis, Postbus 2500, Nieuwegein
  - Multiple Clerosis Center Nijmegen, Heiweg 97, Nyimegen
  - Erasmus MC, Dr. Molewaterplein 40, Rotterdam
  - Sint Elisabeth Ziekenhuis, Hilvarenbeekse Weg 60, Tilburg
  - Maaslandziekenhuis Sittard, Walramstraat 23, BK Sittard
- Poland (10):
  - Samodzielny Publiczny Szpital Kliniczny, Klinika Neurologii, Ul. Marii Skłodowskiej-Curie 24 A, Bialystok
  - Niezalezny Zespol Opieki Zdrowotnej Kendron, Ul. Swietego Mikolaja 1/8, Bialystok
  - Oddzial Neurologiczny i Leczenia Udarow, Mozgu, Nowe Ogrody 1/6, Gdańsk
  - Katedra i Klinika Neurologii Slaskiej Akademii Medycznej, Ul. Medykow 14, Katowice
  - Univ. Med. Sci. Poznan, Katedra i Klinika Neurologii,, Department of Neurology, Ul. Przybyszewskiego 49, Poznan
  - CSK MSWiA Hospital, Department of Neurology, Wołoska 137, Warsaw
  - Jadwiga Kruszewska-Ozimska, Instytut Psychiatrii i Neurologii, II Klinika Neurologii, Ul. Sobieskiego 1/9, Warsaw
  - Centralny Szpital Kliniczny, Klinika Neurologii, MSWiAw Warszawie, Woloska 137, Warszawa
  - Katedra i Klinika Neurologii Centralny Szpital Kliniczny AM w Warszawie, Ul. Banacha 1A, Warszawa
  - Medical University of Lodz, Lodz
- Russia (5):
  - Interregional Clinical Diagnistic Center, Neurology Department, Kazan'
  - Central Clinical Hospital of Medical Center of Administration of President of Russian Federation, Moscow
  - Moscow Regional Research Clinical Institue, Moscow
  - Military Medical Academy, Neurology Department, Saint Petersburg
  - GUZ "Central Medical Sanitary Department #122 of Federal Medical-Biological agency", Neurology department, Saint Petersburg
- Slovakia (4):
  - II. Neurologická klinika Fakultná nemocnica s poliklinikou Bratislava pracovisko Kramáre, Limbová 5, Bratislava Region
  - Neurologická klinika, Martinská fakultná nemocnica, Kollárova 2, Martin
  - I. Neurologická klinika, Fakultná nemocnica s poliklinikou Bratislava pracovisko Staré mesto, Mickiewiczova 13, Bratislava
  - Neurologické oddelenie, Nemocnica s poliklinikou Žilina, ul.V. Spanyola 43, Žilina
- South Africa (3):
  - Umhlanga Hospital, Umhlanga, KwaZulu-Natal
  - Division of Neurology, Groote Schuur Hospital, E 8-74, Groote Schuur Hospital, Observatory Cape Town
  - Private Neurologist (Morningside Medi-Clinic), Suite C, Block C, Rochester Place, Sandton
- Sweden (3):
  - MS Centrum, Forskningsenhet, SU/Östra CKÖ Plan 0, Gothenburg
  - Karolinska University Hospital Huddinge, Department of Neurology R54, Stockholm
  - Karolinska University Hospital, Department of Medicine, Neuroimmunology Unit, CMM L8:04, Stockholm
- Switzerland (3):
  - Kantonsspital Basel, Policlinic, Neurology-Neurosurgical, Petersgraben 4, Basel
  - Centre Hospitalier, Universitaire Vaudois Policlinique de Neurologie, Rue Du Bugnon, Lausanne
  - UniversitätsSpital Zürich, Neurologische Klinik, Frauenklinikstr. 26, Zurich
- Turkey (Türkiye) (12):
  - Hacettepe Universiti Hospitals, Department of Neurology, Ankara
  - Gazi University, Medical Faculty Neurology Department, Besevler Ankara
  - EGE University, Medical Faculty Hospital Neurolgy Department, Bornova Izmir
  - Istanbul University, Istanbul Faculty of Medicine, Departement of Neurology, Capa Istanbul
  - Istanbul University, Cerrahpasa School of Medicine, Department of Neurology, Cerrahpasa Istanbul
  - Gaziantep University School of Medicine, Neurology Department, Gaziantep
  - Uludag University Faculty of Medche, Tip Fakultesi, Noroloji ABD, Görükle / Bursa
  - Tepecik Training and Research, Hospital Neurology Service, 35120 Gaziler Cad. Izmir
  - Dokuz University Medical Faculty, Neurology Department, Inciralti, Izmir
  - Bakirkoy Ruh ve Sinir Hastaliklari Hastanesi, Istanbul
  - Mersin Universitesi Tip Fakultesi Hastanesi, Noroloji ABD, Mersin
  - T.C. Saglik Bakanligi Goztepe Egitim ve Arastirma Hastanesi, Noroloji Klinigi, Göztepe Istanbul
- United Kingdom (6):
  - King's College Hospital, Trials office Academie Neuroscience Center, P041 Institute of Psychiatry, Denmark Hill, London
  - Queens Medical Centre, Division of Clinical Neurology Medical School, Nottingham
  - Royal Hallamshire Hospital, Glossop Road, Sheffield
  - St. George's Hospital, Neurology Dept. Atkinson Morley Wing, Backshaw Road, London
  - Frenchay Hospital, Department of Neurology, Beckspool Road, Bristol
  - Royal Victoria Infirmary, Queen Victoria Road, Newcastle-upon-Tyne

REFERENCES:
- [Derived] Nowak CP, Mutze T, Konietschke F. Group sequential methods for the Mann-Whitney parameter. Stat Methods Med Res. 2022 Oct;31(10):2004-2020. doi: 10.1177/09622802221107103. Epub 2022 Jun 13. PMID 35698787
- [Derived] Fox RJ, Chan A, Zhang A, Xiao J, Levison D, Lewin JB, Edwards MR, Marantz JL. Comparative effectiveness using a matching-adjusted indirect comparison between delayed-release dimethyl fumarate and fingolimod for the treatment of multiple sclerosis. Curr Med Res Opin. 2017 Feb;33(2):175-183. doi: 10.1080/03007995.2016.1248380. Epub 2016 Nov 10. PMID 27733070
- [Derived] Derfuss T, Bergvall NK, Sfikas N, Tomic DL. Efficacy of fingolimod in patients with highly active relapsing-remitting multiple sclerosis. Curr Med Res Opin. 2015;31(9):1687-91. doi: 10.1185/03007995.2015.1067191. Epub 2015 Aug 20. PMID 26121423
- [Derived] Kremenchutzky M, O'Connor P, Hohlfeld R, Zhang-Auberson L, von Rosenstiel P, Meng X, Grinspan A, Hashmonay R, Kappos L. Impact of prior treatment status and reasons for discontinuation on the efficacy and safety of fingolimod: Subgroup analyses of the Fingolimod Research Evaluating Effects of Daily Oral Therapy in Multiple Sclerosis (FREEDOMS) study. Mult Scler Relat Disord. 2014 May;3(3):341-9. doi: 10.1016/j.msard.2013.10.006. Epub 2013 Nov 5. PMID 25876471
- [Derived] Chinea Martinez AR, Correale J, Coyle PK, Meng X, Tenenbaum N. Efficacy and safety of fingolimod in Hispanic patients with multiple sclerosis: pooled clinical trial analyses. Adv Ther. 2014 Oct;31(10):1072-81. doi: 10.1007/s12325-014-0154-4. Epub 2014 Sep 23. PMID 25245812
- [Derived] Zarbin MA, Jampol LM, Jager RD, Reder AT, Francis G, Collins W, Tang D, Zhang X. Ophthalmic evaluations in clinical studies of fingolimod (FTY720) in multiple sclerosis. Ophthalmology. 2013 Jul;120(7):1432-9. doi: 10.1016/j.ophtha.2012.12.040. Epub 2013 Mar 24. PMID 23531349
- [Derived] Radue EW, O'Connor P, Polman CH, Hohlfeld R, Calabresi P, Selmaj K, Mueller-Lenke N, Agoropoulou C, Holdbrook F, de Vera A, Zhang-Auberson L, Francis G, Burtin P, Kappos L; FTY720 Research Evaluating Effects of Daily Oral Therapy in Multiple Sclerosis (FREEDOMS) Study Group. Impact of fingolimod therapy on magnetic resonance imaging outcomes in patients with multiple sclerosis. Arch Neurol. 2012 Oct;69(10):1259-69. doi: 10.1001/archneurol.2012.1051. PMID 22751847
- [Derived] Devonshire V, Havrdova E, Radue EW, O'Connor P, Zhang-Auberson L, Agoropoulou C, Haring DA, Francis G, Kappos L; FREEDOMS study group. Relapse and disability outcomes in patients with multiple sclerosis treated with fingolimod: subgroup analyses of the double-blind, randomised, placebo-controlled FREEDOMS study. Lancet Neurol. 2012 May;11(5):420-8. doi: 10.1016/S1474-4422(12)70056-X. Epub 2012 Apr 10. PMID 22494956
- [Derived] Kappos L, Radue EW, O'Connor P, Polman C, Hohlfeld R, Calabresi P, Selmaj K, Agoropoulou C, Leyk M, Zhang-Auberson L, Burtin P; FREEDOMS Study Group. A placebo-controlled trial of oral fingolimod in relapsing multiple sclerosis. N Engl J Med. 2010 Feb 4;362(5):387-401. doi: 10.1056/NEJMoa0909494. Epub 2010 Jan 20. PMID 20089952
- See also: Fingolimod clinical trials information website — http://www.msclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Started | 429 | 425 | 418
Completed | 332 (296 completed on study drug, 35 completed off study drug.) | 369 (345 completed on study drug, 24 completed off study drug.) | 332 (303 completed on study drug, 29 completed off study drug.)
Not Completed | 97 | 56 | 86
Not completed — Withdrawal by Subject | 31 | 17 | 28
Not completed — Adverse Event | 22 | 13 | 18
Not completed — Lack of Efficacy | 13 | 6 | 25
Not completed — Abnormal laboratory value(s) | 20 | 9 | 1
Not completed — Lost to Follow-up | 3 | 5 | 7
Not completed — Protocol Violation | 5 | 5 | 4
Not completed — Abnormal test procedure result(s) | 2 | 1 | 1
Not completed — Death | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo | Total
Number analyzed (Participants) | 429 | 425 | 418 | 1272
Age Continuous [Mean (Standard Deviation); unit: years] | 37.4 (8.91) | 36.6 (8.77) | 37.2 (8.60) | 37.1 (8.76)
Age, Customized [Number; unit: participants]
  <18 years | 1 | 0 | 0 | 1
  18 -30 | 107 | 120 | 97 | 324
  31-40 | 147 | 162 | 165 | 474
  41-55 | 174 | 143 | 156 | 473
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 295 | 296 | 298 | 889
  Male | 134 | 129 | 120 | 383
Duration of multiple sclerosis since first symptoms [Mean (Standard Deviation); unit: Years] | 8.4 (6.86) [0 to 37] | 8.0 (6.60) [0 to 35] | 8.1 (6.35) [0 to 32] | 8.2 (6.60) [0 to 37]
Number of relapses in last 2 years [Mean (Standard Deviation); unit: relapses] | 1.5 (0.81) [1 to 10] | 1.5 (0.76) [1 to 11] | 1.4 (0.73) [1 to 10] | 1.5 (0.77) [1 to 11]
Expanded Disability Status Scale (EDSS) [Mean (Standard Deviation); unit: Units on a scale] — The EDSS is a scale for assessing disability in 8 functional systems (visual, brain stem, pyramidal, cerebellar, sensory, bowel & bladder, cerebral, other functions). Based on scores in these 8 functional systems, an overall score ranging from 0 (normal) to 10 (death due to MS) is assigned. Patients with EDSS scores of 0.0 to 4.5 are fully ambulatory; patients with EDSS scores of 5.0 to 9.5 have impaired ambulation. EDSS was assessed by an evaluating physician at each site.
  Units on a scale | 2.41 (1.36) [0 to 5.5] | 2.30 (1.29) [0 to 5.5] | 2.49 (1.29) [0 to 5.5] | 2.40 (1.32) [0 to 5.5]

OUTCOME MEASURES:

1. Primary Outcome: Estimated Annualized Aggregate Relapse Rate (ARR)
Description: The ARR is defined as the number of confirmed relapses in a year. A relapse is defined as the appearance of a new or worsening of a previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding relapse. The abnormality must be present for at least 24 hours and occur in the absence of fever or infection. The annualized ARR for each treatment group was the mean of the annualized ARRs for all patients in the group calculated as the total number of confirmed relapses divided by the total number of days on study, multiplied by 365.25.
Time Frame: Baseline to end of study (Month 24)
Population: This analysis was conducted using the Intent-to-treat (ITT) population which includes all patients who were randomized and received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Relapses per year
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 429 | 425 | 418
Relapses per year | 0.16 [0.13 to 0.19] | 0.18 [0.15 to 0.22] | 0.40 [0.34 to 0.47]

2. Secondary Outcome: Percentage of Patients Free of Disability Progression at Month 24 Assessed With the Expanded Disability Status Scale (EDSS)
Description: EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) is calculated. Disability progression was determined by the following: One point increase from baseline in patients with baseline EDSS score from 0 to 5.0; or half a point increase in patients with baseline EDSS score of 5.5 or above. A 3-month confirmed disability progression required onset EDSS, 3-month confirming EDSS, and all EDSS in between to meet the disability progression criteria. Percent of free of disability progression was calculated using the Kaplan Meier method.
Time Frame: Baseline to end of study (Month 24)
Population: Intent-to-treat population (ITT): All patients who were randomized and received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 429 | 425 | 418
Percentage of participants | 83.4 (1.87) [79.7 to 87.1] | 82.3 (1.89) [78.6 to 86.1] | 75.9 (2.17) [71.7 to 80.2]

3. Secondary Outcome: Number of New or Newly Enlarged T2 Lesions at Month 24 in Comparison With Baseline
Description: The number of new or newly enlarged T2 lesions at Month 24 in comparison to baseline was assessed with T2-weighted magnetic resonance image (MRI) scans. A T2-weighted MRI scan utilizes particular values of the echo time (TE) and the repetition time (TR) parameters of image acquisition. Inflammation and tissue damage are seen as bright areas in T2 images and are often referred to as T2 lesions. T2-weighted MRI scans are a sensitive way to evaluate the brain for demyelinating diseases, such as multiple sclerosis.
Time Frame: Baseline to end of study (Month 24)
Population: Intent-to-treat population (ITT): All patients who were randomized and received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: T2 lesions
Units Other Than Participants: patients with non-missing values
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Number analyzed (Participants) | 429 | 425 | 418
Number analyzed (patients with non-missing values) | 337 | 370 | 339
T2 lesions | 2.5 (5.52) | 2.5 (7.19) | 9.8 (13.17)

ADVERSE EVENTS:
Time Frame: 24 Months
Description: Adverse events are reported based on the safety population. The safety population consists of all patients who received at least 1 dose of study drug.
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 51/429 | 43/425 | 56/418
Other Adverse Events (participants affected / at risk) | 346/429 | 355/425 | 323/418
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 1.25 mg (N=429) | Fingolimod 0.5 mg (N=425) | Placebo (N=418)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 3 | 4 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 1
Macular oedema (Eye disorders) | 3 | 0 | 0
Papilloedema (Eye disorders) | 1 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Retinal disorder (Eye disorders) | 1 | 0 | 0
Retinitis (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Chest pain (General disorders) | 0 | 2 | 0
Fatigue (General disorders) | 1 | 0 | 0
Haemorrhagic cyst (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Abscess (Infections and infestations) | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0
Dermo-hypodermitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Genital herpes (Infections and infestations) | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0
Peritoneal abscess (Infections and infestations) | 0 | 0 | 1
Peritonsillitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Streptococcal abscess (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Electrocardiogram PR prolongation (Investigations) | 1 | 0 | 0
Electrocardiogram change (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 2 | 0 | 1
Precancerous cells present (Investigations) | 1 | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 2
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 2 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 1 | 0
Monoplegia (Nervous system disorders) | 0 | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 2 | 0
Multiple sclerosis relapse (Nervous system disorders) | 3 | 2 | 1
Partial seizures with secondary generalisation (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 3
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 2 | 0 | 1
Homicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 1.25 mg (N=429) | Fingolimod 0.5 mg (N=425) | Placebo (N=418)
Vertigo (Ear and labyrinth disorders) | 18 | 18 | 21
Diarrhoea (Gastrointestinal disorders) | 40 | 50 | 30
Nausea (Gastrointestinal disorders) | 38 | 38 | 36
Fatigue (General disorders) | 46 | 48 | 45
Bronchitis (Infections and infestations) | 39 | 34 | 15
Influenza (Infections and infestations) | 40 | 55 | 41
Nasopharyngitis (Infections and infestations) | 112 | 115 | 115
Pharyngitis (Infections and infestations) | 25 | 26 | 23
Rhinitis (Infections and infestations) | 18 | 25 | 25
Sinusitis (Infections and infestations) | 27 | 27 | 19
Upper respiratory tract infection (Infections and infestations) | 62 | 73 | 72
Urinary tract infection (Infections and infestations) | 21 | 34 | 47
Alanine aminotransferase increased (Investigations) | 49 | 42 | 16
Gamma-glutamyltransferase increased (Investigations) | 31 | 22 | 4
Weight increased (Investigations) | 14 | 14 | 22
Hypercholesterolaemia (Metabolism and nutrition disorders) | 26 | 24 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 30 | 33
Back pain (Musculoskeletal and connective tissue disorders) | 45 | 49 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 28 | 27
Dizziness (Nervous system disorders) | 31 | 31 | 23
Headache (Nervous system disorders) | 113 | 107 | 96
Paraesthesia (Nervous system disorders) | 17 | 23 | 18
Depression (Psychiatric disorders) | 25 | 33 | 28
Insomnia (Psychiatric disorders) | 16 | 21 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 43 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 30 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 29 | 29
Hypertension (Vascular disorders) | 27 | 26 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.